CLINICAL TRIAL: NCT05973968
Title: A Real-world Study of Surufatinib in Refractory Metastatic G3 Neuroendocrine Tumors
Brief Title: Surufatinib in G3 Neuroendocrine Tumors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); The Affiliated Hospital of Qingdao University (Other); Yantai Yuhuangding Hospital (Other); Weifang People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202210-028-1
Record Dates: First submitted 2023-07-16; First posted 2023-08-03 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-04

CONDITIONS: Neuroendocrine Tumor Grade 3
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surufatinib: Surufatinib 300mg QD, po, every 4 weeks as a course of treatment, continuous administration until PD, death or intolerable toxicity
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Taking 28 days as a treatment cycle, the tumor was evaluated by imaging method every 8 weeks (±7 days) in the first 52 weeks, and then every 12 weeks (±7 days) until the disease progression (RECIST1.1) or death (during the treatment of the patient). The treatment and survival status of the tumor after disease progression were recorded.

SUMMARY:
The goal of this observational study is to learn about surufatinib in Refractory Metastatic G3 Neuroendocrine Tumors. The main questions it aims to answer are:

* To evaluate the efficacy and safety of surufatinib in the treatment of second-line and posterior-line in G3 neuroendocrine tumors.
* To explore the predictive value of blood perfusion parameters in curative effect.

Participants will be given surufatinib 300mg QD, po, every 4 weeks as a course of treatment, continuous administration until PD, death or intolerable toxicity.

DETAILED DESCRIPTION:
Currently, there is a lack of standard treatment for metastatic G3 neuroendocrine tumors, and CSCO guidelines recommend patients to enter clinical trials. The NCCN guidelines recommend that patients with G3 be divided into two groups according to Ki67 > 55%, SSTR expression, tumor load and progression, and are treated with chemotherapy, somatostatin, mTOR inhibitor, and Sunitinib (limited to pancreatic neuroendocrine tumors). Among them, a small sample study showed that there was no significant difference in the efficacy of sunitinib in the treatment of pancreatic neuroendocrine tumors (PFS) between G3 and G1/2.

surufatinib capsule is a new oral tyrosine kinase inhibitor. Approved by NMPA for unresectable locally advanced or metastatic, advanced non-functional, well differentiated (G1, G2) non-pancreatic (December 2020) and pancreatic (June 2021) neuroendocrine tumors, in the 2022 Chinese guidelines for integrated diagnosis and treatment of tumors, it is recommended to choose surufatinib after the second line of treatment for G3 NEN patients with Ki67 < 55%. However, there is still a lack of data on the efficacy and safety of surufatinib in the real world in China, and its efficiency in G3 NEN is worth exploring.

The goal of this observational study is to learn about surufatinib in Refractory Metastatic G3 Neuroendocrine Tumors. The main questions it aims to answer are:

* To evaluate the efficacy and safety of surufatinib in the treatment of second-line and posterior-line in G3 neuroendocrine tumors.
* To explore the predictive value of blood perfusion parameters in curative effect.

Participants will be given surufatinib 300mg QD, po, every 4 weeks as a course of treatment, continuous administration until PD, death or intolerable toxicity.

Taking 28 days as a treatment cycle, the tumor was evaluated by imaging method every 8 weeks (±7 days) in the first 52 weeks, and then every 12 weeks (±7 days) until the disease progression (RECIST1.1) or death (during the treatment of the patient). The treatment and survival status of the tumor after disease progression were recorded.

Safety indicators include: adverse events, laboratory tests, vital signs and changes in ECG and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood this study and voluntarily signed the informed consent form;
2. Age ≥ 18 years old, both male and female;
3. Neuroendocrine tumors diagnosed by histopathology or cytology (patients with neuroendocrine tumors diagnosed as G3 according to WHO2019 criteria, and Ki67 index ≤ 55%);
4. Progress after at least one systemic chemotherapy;
5. According to the evaluation criteria of solid tumor efficacy (RECISTV1.1), there is at least one measurable lesion.
6. Palliative radiotherapy at the localized site was allowed for more than 7 days since the end of the last systematic treatment, which has been over 4 weeks.
7. Expected survival ≥ 12 weeks;
8. The researchers assessed that they could benefit;
9. Have enough organ and bone marrow function;
10. Fertile male or female patients voluntarily used effective contraceptive methods during the study period and within 6 months of the last study, such as double barrier contraceptives, condoms, oral or injection contraceptives, intrauterine devices, etc. All female patients will be considered fertile unless the female patient has undergone natural menopause, artificial menopause or sterilization (such as hysterectomy, bilateral adnexectomy or radioactive ovarian irradiation). Otherwise, the serum of female patients showed that they were not pregnant within 7 days before the study and must be non-lactation patients.

Exclusion Criteria:

1. Other malignant tumors have been diagnosed in the past 5 years, except for skin basal cell carcinoma, skin squamous cell carcinoma, cervical cancer in situ and breast cancer after effective treatment.
2. At the same time, receive other experimental drugs or approved or under research anti-tumor therapy;
3. Patients with contraindications of Surufatinib (such as active bleeding, ulcer, intestinal perforation, intestinal obstruction, uncontrollable hypertension, III-IV cardiac insufficiency, severe hepatic and renal insufficiency within 30 days after major operation, etc.).
4. The patient currently has any disease or condition that affects drug absorption, or the patient cannot take Surufatinib orally;
5. It has been proved to be allergic to experimental drugs and any components in their excipients;
6. Women who are pregnant (positive for pre-medication pregnancy test) or breastfeeding;
7. Patients with large pleural effusion or ascites need drainage;
8. Any other disease, with clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the researchers, there is reason to suspect that the patient has a disease or state that is not suitable for the use of research drugs (such as having seizures and requiring treatment), or will affect the interpretation of the findings or put the patient at high risk;
9. Drugs containing Hypericum perforatum were taken within 3 weeks before treatment, or other strong inducers or inhibitors of CYP3A4 were taken in the previous 2 weeks.
10. According to the researchers, the subjects have other factors that may lead to the termination of this study or are not suitable for inclusion, such as other serious concomitant diseases (such as severe diabetes, thyroid disease, spinal cord compression, superior vena cava syndrome, mental illness), severe laboratory abnormalities, family or social factors, which will affect the safety of the subjects, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with G3 neuroendocrine tumor
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | through study completion, an average of 1 year
  Progression Free Survival

SECONDARY OUTCOMES:
objective response rate | through study completion, an average of 1 year
  objective response rate
overall survival | through study completion, an average of 1 year
  overall survival
disease control rate | through study completion, an average of 1 year
  disease control rate
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 1 year
  Including type, incidence, grading (according to NCI-CTCAEV5.0), severity.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hofland J, Kaltsas G, de Herder WW. Advances in the Diagnosis and Management of Well-Differentiated Neuroendocrine Neoplasms. Endocr Rev. 2020 Apr 1;41(2):371-403. doi: 10.1210/endrev/bnz004. PMID 31555796
- [Result] Raymond E, Dahan L, Raoul JL, Bang YJ, Borbath I, Lombard-Bohas C, Valle J, Metrakos P, Smith D, Vinik A, Chen JS, Horsch D, Hammel P, Wiedenmann B, Van Cutsem E, Patyna S, Lu DR, Blanckmeister C, Chao R, Ruszniewski P. Sunitinib malate for the treatment of pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):501-13. doi: 10.1056/NEJMoa1003825. PMID 21306237
- [Result] Yao JC, Fazio N, Singh S, Buzzoni R, Carnaghi C, Wolin E, Tomasek J, Raderer M, Lahner H, Voi M, Pacaud LB, Rouyrre N, Sachs C, Valle JW, Fave GD, Van Cutsem E, Tesselaar M, Shimada Y, Oh DY, Strosberg J, Kulke MH, Pavel ME; RAD001 in Advanced Neuroendocrine Tumours, Fourth Trial (RADIANT-4) Study Group. Everolimus for the treatment of advanced, non-functional neuroendocrine tumours of the lung or gastrointestinal tract (RADIANT-4): a randomised, placebo-controlled, phase 3 study. Lancet. 2016 Mar 5;387(10022):968-977. doi: 10.1016/S0140-6736(15)00817-X. Epub 2015 Dec 17. PMID 26703889
- [Result] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057
- [Result] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687